CLINICAL TRIAL: NCT02988180
Title: Developmental and Growth Status of Children (6-60 Months of Age) in Extreme Poverty in Jimma Town of Ethiopia: Effects of Developmental Stimulation - RAI (Risk Analysis and Intervention)
Brief Title: Intervention on Development and Growth at Children in Poverty
Acronym: RAI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Collaborators: Jimma University (Other); VLIR-UOS (Vlaamse Interuniversitaire Raad). (Unknown)
Responsible Party: Principal Investigator, prof. dr. Marita Granitzer, prof.dr., Hasselt University
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: DGSC-2015
Record Dates: First submitted 2016-11-17; First posted 2016-12-09 (Estimated); Last update posted 2016-12-09 (Estimated); Status verified 2016-12

CONDITIONS: Child Malnutrition
MeSH Terms: conditions — Child Nutrition Disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- intervention group (Other): Children in the intervention group received basic services such as family-home, food, clothing, health care, protection and education for older children. In addition, there received play-based developmental stimulation integrated into the services.
  Interventions: Other: basic services; Other: the play-based developmental stimulation
- control group (Other): The age-matched control children received the basic services such as family-home, food, clothing, health care, protection and education. However, they were not provided with the play-based developmental stimulation.
  Interventions: Other: basic services

INTERVENTIONS:
Other: basic services — The age-matched control children received the basic services such as family-home, food, clothing, health care, protection and education. However, they were not provided with the play-based developmental stimulation.
Other: the play-based developmental stimulation — Children in the intervention group received basic services such as family-home, food, clothing, health care, protection and education for older children. In addition, there received play-based developmental stimulation integrated into the services.
  Arms: intervention group

SUMMARY:
Children in extreme poverty lack adequate care and face increased health risks. The earlier poverty strikes in the developmental process, the more deleterious and long-lasting its effects. There is, however, growing evidence that early interventions can prevent the negative consequences. Such interventions are effective, particularly when they are of high quality, organized at home and parents are involved. Recently, baseline assessment of developmental and nutritional status of SOS children and children in extreme poverty in Jimma region of South-West Ethiopia revealed that these children have developmental problems in language, motor, social-emotional skills and nutritional status. The impact of play-oriented stimulation activities integrated into the existing SOS basic program, on developmental outcomes, has never been investigated in this context. The main objective of the study is, therefore, to evaluate the impact of play-oriented stimulation integrated into the basic SOS program on the developmental outcomes of children living with foster families. This was done by comparing the intervention children with their age-matched children (control), not receiving the stimulation package. It was hypothesized that this package would significantly improve the developmental skills of these children.

ELIGIBILITY:
Inclusion Criteria:

* Children who were selected by the SOS children's village as lacking parental care and receive basic services;
* Children living in Jimma town;
* Children from 3 months to 59 months of age.

Exclusion Criteria:

* Children with observable physical disabilities which hinders mobility;
* Children with severe mental retardation;
* Children with discernable hearing and visual impairments.

Ages: 3 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 78 (Actual)
Dates: Start 2015-10; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Personal-social outcome | baseline
  Denver II-Jimma was used to test personal-social outcome and performance ratio was calculated for analysis
Personal-social outcome | month 3
  Denver II-Jimma was used to test personal-social outcome and performance ratio was calculated for analysis
Personal-social outcome | month 6
  Denver II-Jimma was used to test personal-social outcome and performance ratio was calculated for analysis
fine motor outcome | baseline
  Denver II-Jimma was used to test fine motor outcome and performance ratio was calculated for analysis
fine motor outcome | 3 months
  Denver II-Jimma was used to test fine motor outcome and performance ratio was calculated for analysis
fine motor outcome | 6 months
  Denver II-Jimma was used to test fine motor outcome and performance ratio was calculated for analysis
gross motor outcome | baseline
  Denver II-Jimma was used to test gross motor outcome and performance ratio was calculated for analysis
gross motor outcome | 3 months
  Denver II-Jimma was used to test gross motor outcome and performance ratio was calculated for analysis
gross motor outcome | 6 months
  Denver II-Jimma was used to test gross motor outcome and performance ratio was calculated for analysis
language outcome | baseline
  Denver II-Jimma was used to test language outcome and performance ratio was calculated for analysis
language outcome | 3 months
  Denver II-Jimma was used to test language outcome and performance ratio was calculated for analysis
language outcoome | 6 months
  Denver II-Jimma was used to test language outcome and performance ratio was calculated for analysis
Social-emotional outcome | baseline
  Ages and Stages Questionnaires: Social Emotional (ASQ: SE) was used to measure social-emotional development of the children
Social-emotional outcome | 3 months
  Ages and Stages Questionnaires: Social Emotional (ASQ: SE) was used to measure social-emotional development of the children
Social-emotional outcome | 6 months
  Ages and Stages Questionnaires: Social Emotional (ASQ: SE) was used to measure social-emotional development of the children

SECONDARY OUTCOMES:
weight | baseline
  A child's weight was measured by using a calibrated electronic weighing scale.
weight | 3 months
  A child's weight was measured by using a calibrated electronic weighing scale.
weight | 6 months
  A child's weight was measured by using a calibrated electronic weighing scale.
Height | baseline
  For children under two years of age, a length measuring board on a flat table was used. For children under two years of age, a length measuring board on a flat table was used. The height of a child above two years of age was measured by using a portable stadiometer.
Height | 3 months
  For children under two years of age, a length measuring board on a flat table was used. The height of a child above two years of age was measured by using a portable stadiometer.
Height | 6 months
  For children under two years of age, a length measuring board on a flat table was used. The height of a child above two years of age was measured by using a portable stadiometer.

CONTACTS AND LOCATIONS:
Overall Officials: Teklu Gemechu Abessa, Study Chair — Jimma University; Mekitie Wondafrash, nutritionist, Study Chair — Jimma University; Patrick Kolsteren, prof.dr, Study Chair — University Ghent; Berhanu Nigussie Worku, psychologist, Study Chair — Jimma University
Locations (2):
- Ghent University, Ghent, Belgium
- 2. Jimma University, Jimma, Ethiopia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Worku BN, Abessa TG, Wondafrash M, Lemmens J, Valy J, Bruckers L, Kolsteren P, Granitzer M. Effects of home-based play-assisted stimulation on developmental performances of children living in extreme poverty: a randomized single-blind controlled trial. BMC Pediatr. 2018 Feb 5;18(1):29. doi: 10.1186/s12887-018-1023-0. PMID 29402258